CLINICAL TRIAL: NCT06043102
Title: A 7 Week, Open Label, Study Evaluating the Efficacy and Safety of TheraClearX on Mitigating Mild to Moderate Acne in Healthy Teenagers and Young Adults
Brief Title: Study Evaluating the Efficacy and Safety of TheraClearX on Mitigating Mild to Moderate Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: Strata Skin Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSKN-TCX-01
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-09

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Open label study evaluating the efficacy and safety
Masking Description: Open label study evaluating the efficacy and safety
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TheraClearX treatment (Other): TheraClearX treatment of the facial area weekly for 6 sessions.
  Interventions: Device: TheraClearX

INTERVENTIONS:
Device: TheraClearX — TheraClear®X combines vacuum pressure with a broadband light source (500 nm to 1,200 nm) to treat facial acne.

SUMMARY:
The goal of this clinical trial is to further substantiate the effectiveness and safety of TheraClearX as a stand-alone treatment of mild to moderate acne in healthy teenagers and adults ages 12-40 over the course of 7 weeks. Participants will be asked to have TheraClearX treatments weekly for 6 sessions, attend a follow up appointment 2 weeks after the 6th session, have photos taken of their face and answer questionnaires related to their acne.

DETAILED DESCRIPTION:
Acne is a common disease of the pilosebaceous unit affecting both teenagers and young adults that causes both physical and emotional damage. The risk of delaying treatment is that of scarring which can be devastating for patients of all ages. The pathogenesis is complex and appears to involve 4 primary features: increased stimulation of sebum gland activity, increased bacterial proliferation (especially Propionibacterium acnes), abnormal follicular hyperkeratinization and resultant obstruction of the sebaceous follicles, and the release of inflammatory mediators. These changes in acne patients result in the formation of clinical inflammatory lesions including superficial pustules such as comedones (popularly known as "blackheads" or "whiteheads") and more deeply located pustules, papules, nodules and cysts.

Due to the complexity of pathogenic mechanisms causing acne, treatment typically includes combination therapy including topical applications, oral medications, and numerous alternative therapies including lasers, light, steroid injections, chemical peels, and extractions. Many of these treatments while effective if used for a sustained period of time, have side effects, complications, and resistance. So it is important to consider alternative therapeutic options. The application of lasers and light-based systems in the field of dermatology has dramatically advanced based on Anderson and Parish's theory of selective photothermolysis in which very short pulses of laser energy with high peak powers at a given wavelength are selectively absorbed by target chromophores such as melanin and hemoglobin, but delivering minimum damage to the normal tissue surrounding the target. The application of these lasers in the extended theory of photothermolysis has currently expanded to include the treatment of acne.

Recently, a novel device called TheraClear®X, that combines vacuum pressure with a broadband light source (500 nm to 1,200 nm) was developed for the treatment of acne. Unlike currently available devices, TheraClear®X uses gentle pneumatic energy to draw the target tissue into the treatment tip, with negative pressure lifting the sebaceous gland and thus bringing it closer to the surface of the skin. The vacuum then elevates and everts the sebaceous gland, allowing it to open up and empty its contents, ejecting the acne causing bacteria, sebum, dead skin cells, and other impurities onto the surface of the skin. Such photopneumatic devices are the only pulsed broadband light therapy approved by the United States Food and Drug Administration for the treatment of comedonal and pustular acne, as well as inflammatory acne. Inflammation caused by acne also has a major vascular component, which appears as redness. Pulsed light is an ideal energy source to remove this redness. Being able to offer comfortable, low risk treatment options for patients suffering with acne is critical as more patients are looking for these options. This clinical trial is therefore a critical addition to the armamentarium of acne treatments. The proposed clinical study will substantiate the efficacy and safety of TheraClear®X as a stand-alone treatment for the mitigation of mild to moderate acne in healthy teenagers and young adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or females of all Fitzpatrick Skin Types between 12 and 40 years of age.
2. Subjects must be willing to provide verbal understanding and sign an Informed Consent Form, HIPAA Form and Photography Release Form approved by the Institutional Review Board. Subjects less than age of consent must sign an assent for the study and a parent must sign the informed consent (if subject reaches the age of consent during the study they should be re-consented at the next study visit).
3. Subjects must be in general good health, as determined by the Investigator.
4. Subjects must be willing and able to attend all study visits and comply with the Pre and Post Treatment Instructions.
5. Subjects must be willing to have VISIA facial photography imaging of their entire face for overall evaluation of their skin at all Visits.
6. Subjects must be willing and able to complete and understand the various rating questionnaires.
7. Subjects must have an IGA score of 2 (mild) or 3 (moderate) at the Baseline Visit.
8. Subjects must have a facial acne inflammatory lesion (papules, pustules, and nodules) count with no less than 10 but no more than 50 at the Baseline Visit.
9. Subjects must have a facial acne non-inflammatory lesion (open and closed comedones) count with no less than 10 but no more than 100 at the Baseline Visit.
10. Subjects with 1 or fewer facial nodules at the Baseline Visit.
11. Females of child bearing potential (FOCBP) and females who are premenses must be willing to practice effective contraception for the duration of the study. (Effective contraception is defined as stabilized on oral contraceptive for at least 3 months, intrauterine device, condom with spermicide, diaphragm with spermicide, implant, NuvaRing®, injection, transdermal patch or abstinence.) Females on birth control pills must have taken the same type pill for at least 3 months prior to entering the study and must not change type during the study. Those who have used birth control pills in the past must have discontinued usage at least 3 months prior to the start of the study. Women who use birth control for acne control only should be excluded.
12. Premenses females and FOCBP must have a negative urine pregnancy test at the Baseline Visit.
13. Subjects must be willing to comply with study instructions and return to the clinic for required visits.
14. Subjects must be willing to use the cleanser, moisturizer and sunscreen provided by the Sponsor.
15. If the subject wears makeup, they must agree to use non-comedogenic makeup.
16. Male subjects facial area must be clean-shaven for all study visits as to not interfere with study treatments and assessments.

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study.
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, Gram- negative folliculitis, dermatitis, eczema.
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
4. Subjects with more than 50 facial acne inflammatory lesions (papules, pustules, and nodules)
5. Subjects with more than 100 facial acne non-inflammatory lesions (open and closed comedones)
6. Subjects with more than one (1) facial nodule.
7. Subjects with a facial beard or mustache that could interfere with the study assessments.
8. Subjects who have a history of experiencing significant burning or stinging when applying any facial treatment (eg, makeup, soap, masks, washes, sunscreens, etc) to their face.
9. Female subjects who are pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study.
10. If female, subject has a history of hirsutism, polycystic ovarian disease or clinically significant menstrual irregularities.
11. Subjects who have a history of light-induced seizures or diseases that may be stimulated by visible light.
12. Subjects currently using photosensitive medications or herbal supplements (ie. Tetracycline and St. John's Wart).
13. Subjects who have a history of blood disorders that alter the ability of blood to coagulate and/or are currently taking anti-coagulants or blood thinning medications.
14. Subjects who have a history of keloid and hypertrophic scar formation.
15. Subjects who have a history of Herpes Simplex in the treatment area, connective tissue damage, immunosuppressive diseases, Systemic Lupus Erythematosus and Porphyria.
16. Subjects who currently have active infections, broken skin, extremely dry skin or open lesions in the treatment area.
17. Treatment of any type of cancer within the last 6 months in the facial area, with the exception of complete surgical excision of skin cancer outside the treatment area.
18. Subjects who have not undergone the specified washout period(s) for the following topical preparations/physical treatments used on the face or subjects who require the concurrent use of any of the following in the treatment area:

    Topical astringents and abrasives on the face 1 week Non-allowed moisturizers or sunscreens on the face 1 week Acne surgery 1 week Antibiotics on the face 2 weeks Other topical anti-acne drugs on the face 2 weeks Soaps containing antimicrobials on the face 2 weeks Light (e.g. LED, PDT) therapy on the face 2 weeks Anti-inflammatory agents and corticosteroids on the face 4 weeks Retinoids, including retinol on the face 4 weeks Chemical peel/Microdermabrasion on the face 4 weeks Laser therapy on the face 4 weeks
19. Subjects who have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications:

    Corticosteroids (including intramuscular injections) (inhaled corticosteroids are allowed) 4 weeks Antibiotics 4 weeks Other systemic acne treatments 4 weeks Systemic retinoids 6 months
20. Subjects who have had Botulinum Toxin or Filler in the facial area in the last 2 weeks or are planning on having Botulinum Toxin or Filler during the duration of the study.
21. Subject intends to use a tanning booth or sunbathe during the study.
22. Subjects who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
23. Subjects with any underlying disease that the investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | Baseline to Day 49 or End of Study (EOS) visit
  Papule - A small, solid elevation less than 5 mm in diameter. Most of the lesion is above the surface of the skin. Pustule - A small circumscribed elevation less than 5 mm in diameter that contains yellow-white exudate.
  Nodule - An inflammatory lesion greater than or equal to 5 mm in diameter.
  Cyst - An inflammatory lesion that contains yellow-white exudate that is greater than or equal to 5mm in diameter.
Change in non-inflammatory lesion counts | Baseline to Day 49 or End of Study (EOS) visit
  Open Comedone - (Black head) A lesion in which the follicle opening is widely dilated with the contents protruding out onto the surface of the skin, with compacted melanin cells giving the plug a black appearance.
  Closed Comedone - (White head) A lesion in which the follicle opening is closed, but the sebaceous gland is enlarged by the pressure of the sebum buildup, which in turn cause the skin around the follicle to thin and become elevated with a white appearance.
Percentage/Proportion of subjects who achieve at least a one-grade reduction in the IGA Score | Baseline to Day 49 or End of Study (EOS) visit
  The Investigator will use the Investigator Global Assessment (IGA) Scale to assess the severity of a subjects' acne. The IGA Scale is a static evaluation of global severity representing clinically meaningful graduations of the disease. The IGA should be performed prior to the lesion count. Subjects are eligible for enrollment if they have facial acne with a global severity grade of a 2 (mild) or a 3 (moderate) on the IGA scale at Baseline. If at Visits Day 7, Day 14, Day 21, Day 28 or Day 35 the subject has an IGA Scale rating of Zero (0)/Clear then the subject will proceed to the EOS Visit two (2) weeks following that Visit and no further TheraClear®X Procedures will be performed.

SECONDARY OUTCOMES:
Improvement in Acne QoL questionnaire scores | Baseline to Day 49 or End of Study (EOS) visit
  The Acne-specific Quality of Life questionnaire (Acne QoL) is a health-related quality of life instrument developed by MERCK & CO., INC. for use in clinical trials to assess the impact of therapy on quality of life among subjects with facial acne. The Acne QoL questionnaire consists of 19 questions. The Acne QoL is self-administrated (i.e. the subject is able to complete the questionnaire without assistance or interpretation from study staff) and should take approximately 10 minutes or less to complete. The scale is called Acne-Specific Quality of Life Questionnaire and the scale goes from 0 (not at all) to 6 (extremely). A decrease in response values (lower scores means a better outcome) at Day 49 or EOS indicates an improvement compared to baseline response values.
Improvement in Acne Self Assessment questionnaire scores | Baseline to Day 49 or End of Study (EOS) visit
  The Acne Self-Assessment Questionnaire will ask subjects a series of questions related to their facial acne and overall facial skin appearance. The scale is called the Acne Self-Assessment quesitonnaire and the scale goes from 0 (Very satisfied) to 5 (Very dissatisfied). A decrease in response values (lower scores means a better outcome) at Day 49 or EOS indicates an improvement compared to baseline response values.
Favorable Analysis of the Acne Subject Satisfaction questionnaire | Day 49 or EOS visit
  The Acne Subject Satisfaction Questionnaire will ask subjects a series of questions related to their opinion of treatment satisfaction. The scale is called the Acne Subject Satisfaction questionnaire and the scale goes from 1 (Very Satisfied) to 5 (Very Dissatisfied). Favorable analysis at Day 49 or EOS would be indicated by low response values.
Favorable Analysis of the Subject Consumer Perception questionnaire | Day 49 or EOS visit
  The Subject Consumer Perception Questionnaire will ask subjects a series of questions related to their opinion of what is important to them when choosing an acne treatment. The scale is called the Subject Consumer Perception questionnaire and the scale goes from 1 (Very Likely) to 5 (Very Unlikely). Favorable analysis at Day 49 or EOS would be indicated by low response values.

OTHER OUTCOMES:
Improvement in the VISIA photography imaging of the left, right and front views of the face. | Baseline to Day 49 or EOS visit
  Subjects will have VISIA Facial imaging photographs taken of the right, central and left views of the face prior to TheraClear®X treatment. All VISIA facial images (Standard, Cross-Polarized and UV) will be analyzed to acquire the following data points: (1) SPOTS (2) WRINKLES (3) TEXTURE (4) PORES (5) UV SPOTS (6) BROWN SPOTS (7) RED AREAS (8) PORPHYRINS The VISIA software also formulates the following Ratings for Spots, Wrinkles, Texture, Pores, UV Spots, Brown Spots, Red Areas and Porphyrins: (1) PERCENTILE - This compares the subject to people their same age and their skin type therefore the higher the percentile score the better (2) SCORE - This is the area score that tells how much space the feature is taking up inside the mask therefore the lower the area score the better since this shows when the feature starts to shrink and fade away (3) FEATURE COUNT - Feature counts show how many features are counted during analysis therefore the lower the feature count the better.
The frequency of both local and systemic AE's | Baseline, Day 7, Day 14, Day 21, Day 28, Day 35 and Day 49 or End of Study visit.
  An adverse event is any adverse change from the subject's baseline condition, i.e. any subjective signs and symptoms, or change in a concomitant disease present at the screening visit. This includes inter-current signs, symptoms, illness and significant deviations from baseline which may occur during the course of the clinical study, whether considered related to treatment or not.
Investigator Tolerability Assessment (erythema, edema, dryness, scaling, hypopigmentation and hyperpigmentation) | Baseline, Day 7, Day 14, Day 21, Day 28, Day 35 and Day 49 or End of Study visit.
  The scale is called Investigator Tolerability Assessment and the scale is 0 (None) to 3 (Severe). The scale measures erythema, edema, dryness, scaling, hypopigmentation and hyperpigmentation. A decrease in scores (lower scores are a better outcome) or lack of significant increase at Day 7, Day 14, Day 21, Day 28, Day 35 and Day 49 or EOS comparison to Baseline indicates tolerability/safety of the test device.
Subject Tolerability Self-Assessment (itching, burning and stinging) | Baseline, Day 7, Day 14, Day 21, Day 28, Day 35 and Day 49 or End of Study visit.
  The scale is called Subject Tolerability Assessment and the scale is 0 (None) to 3 (Severe). The scale measures itching, burning and stinging. A decrease in scores (lower scores are a better outcome) or lack of significant increase at Day 7, Day 14, Day 21, Day 28, Day 35 and Day 49 or EOS comparison to Baseline indicates tolerability/safety of the test device.

CONTACTS AND LOCATIONS:
Locations (1):
- Ablon Skin Institute & Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ablon G. A Seven-week, Open-label Trial Evaluating the Safety and Efficacy of a Photopneumatic Device for Mitigating Mild-to-Moderate Acne in Healthy Adolescents and Young Adults. J Clin Aesthet Dermatol. 2024 Jun;17(6):13-20. PMID 38912192